CLINICAL TRIAL: NCT04511754
Title: Experiential Training in Disclosure Elicitation and Emotional Awareness and Activation: A Randomized Test
Brief Title: Experiential Training in Eliciting Disclosure & Emotions for Mental Health Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mark A. Lumley (Other)
Responsible Party: Sponsor-Investigator, Mark A. Lumley, Distinguished Professor of Psychology, Wayne State University
Organization: Wayne State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB20062468B3
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Trauma; Emotions; Disclosure
Keywords: Clinical Training; Mental Health Trainees; Experiential
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at a 1:1 ratio to either the standard training or the experiential training condition.
Who Masked: Outcomes Assessor
Masking Description: Both trainee and researcher will be blinded to training condition assignment prior to randomization, and follow-up assessment will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiential Training Condition (Experimental): Trainees will be taught the following skills during a single session: 1) Therapist in-session emotional-awareness and self-regulation; 2) Facilitating client disclosure of traumas and other difficult experiences; and 3) Helping clients access and experience adaptive emotions. In the experiential training condition, the trainees will receive information about the skills with examples and will have opportunity to practice using short video clips of actors portraying clients. The trainees will be asked to respond to the short clips using the skills they learned. A trainer (a graduate student in clinical psychology) will pause and process the trainees' reactions after they respond to each practice video clip and will provide feedback to the trainees about their performance on the practice.
  Interventions: Behavioral: Experiential Psychotherapy Skill Training
- Standard Training Condition (Active Comparator): Trainees will be taught the following skills during a single session: 1) Therapist in-session emotional-awareness and self-regulation; 2) Facilitating client disclosure of traumas and other difficult experiences; and 3) Helping clients access and experience adaptive emotions. In the standard training condition, the trainee will receive a lecture about the skills including rationale and research background, examples, and opportunities to ask questions. The standard training condition will not include opportunities for practice or live discussion and feedback from the trainer.
  Interventions: Behavioral: Standard Psychotherapy Skill Training

INTERVENTIONS:
Behavioral: Experiential Psychotherapy Skill Training — The Experiential Training intervention will include components of training not usually included in standard clinical training experiences; such components include opportunities for deliberate practice of the skills trained, live supervision and feedback, and discussion with a trainer focused on the skills taught and the trainees' performance.
  Arms: Experiential Training Condition
Behavioral: Standard Psychotherapy Skill Training — Standard didactic training with research support, examples, and opportunities to ask questions.
  Arms: Standard Training Condition

SUMMARY:
Many people seek psychotherapy to alleviate symptoms related to trauma and stressful conflicts, and many psychotherapy approaches aim to help people process trauma and conflicts through eliciting client disclosure of these experiences and activating related emotions. However, many therapists avoid implementing such approaches because they are emotionally challenging for both the client and the therapist, and because therapists lack direct training in specific skills related to eliciting client disclosure and working with emotions. This suggests that providing therapists with a training experience that is experiential, includes direct supervision and feedback, and addresses therapists' reservations and anxieties may be an important approach to increase therapist skills in disclosure elicitation and emotional activation.

This is a randomized trial that will test two methods of training (experiential vs. standard) of master's level psychotherapy students in specific therapeutic skills aimed at increasing trainees' emotional awareness and self-regulation and reducing trainee anxiety and avoidance of eliciting disclosure and working with emotions in psychotherapy. In the standard training condition, the trainee will receive a lecture about the skills including rationale and research background, examples, and opportunities to ask questions. In the experiential training condition, the trainees will receive information about the skills with examples and will have opportunity to practice using short video clips of actors portraying clients. The trainees will be asked to respond to the short clips using the skills they learned, and a trainer will process the trainees' reactions after they respond to each practice video clip and will provide feedback to the trainees about their performance on the practice. Findings from this study will provide information about the feasibility of training in specific disclosure elicitation and emotional activation therapy skills, and will provide information about whether or not live supervision will lead to greater improvement in the targeted skills compared to entirely standard training.

DETAILED DESCRIPTION:
Experiences of trauma and stressful conflicts are common, with most adults in the United States reporting experiences of at least one traumatic event in their lifetimes. Experiences of stressful events vary, and may include war-related trauma, physical, emotional, and sexual abuse, witnessing violence or substance use in the household, and emotional and physical neglect. Exposure to traumatic and stressful events has been linked to adverse physical and psychological health outcomes, impaired functioning, and substantial reductions in quality of life. In addition to trauma exposure, many individuals experience interpersonal and intrapersonal conflicts such as experiences of social rejection, struggles with intimacy or autonomy in relationships, shameful secrets, and perfectionism. Such conflicts are also associated with poor psychological and physical health outcomes. Experiences of trauma and stressful conflicts often underlie many psychological problems that lead individuals to seek psychotherapy.

Many psychotherapy approaches aim to help people disclose and process difficult experiences and activate and experience their emotions, and research suggests that such psychotherapies improve psychological and physical health. For example, written emotional disclosure (or expressive writing) is a therapeutic approach in which a person is asked to write repeatedly about private stressful experiences and avoided emotions. Another psychotherapy approach, Prolonged Exposure Therapy (PE), is designed to help clients approach feared and avoided trauma-related material including memories, thoughts, emotions, and real-life situations. Short-Term Psychodynamic Psychotherapy (STPP) is an approach that helps clients acknowledge and engage with avoided emotions and psychological conflicts and express blocked emotions. One variant of STPP has been used to specifically treat affect phobia, a phobia of experiencing or expressing certain emotions. Emotional Awareness and Expression Therapy (EAET) borrows from STPP, exposure therapy, expressive writing, and other emotion-focused approaches and aims to help people disclose stressful experiences and emotional conflicts and experience and express their emotions related to stressful situations.

The aforementioned psychotherapy approaches have shown benefits for a range of populations and psychological and physical health outcomes; however, this therapeutic work can be challenging, and therapists may often avoid implementing such approaches and skills. Eliciting client disclosure and emotional activation can be especially challenging for novel therapists who may avoid directly inquiring about clients' traumas and conflicts and may experience difficulty tuning into and working with clients' emotions. These barriers are often observed in the implementation of exposure-based approaches, which are underutilized in day-to-day clinical practice. Barriers to therapist implementation of exposure-based techniques include lack of adequate training, the belief that exposure is likely to lead to an increase in symptoms or problems in therapy, and lack confidence in one's ability to handle a range of client emotional reactions.

Comprehensive training experiences are needed to address therapist-centric barriers to utilization of disclosure elicitation and emotional activation skills and to increase therapist self-efficacy related to such skills. Research suggests that entirely didactic training methods, such as reading manuals or watching lectures and training videos, are insufficient to lead to therapist behavior change. Several studies have highlighted the importance of supervision and supervisor feedback in increasing therapist knowledge, proficiency, and retention of therapeutic skills. Additionally, some researchers have highlighted the importance of key components of skill acquisition, such as repetitive or deliberate practice of specific skills through role plays and simulations, personalized performance feedback, and experiential/reflective training approaches. Therapist self-reflection and self-regulation practices have also been highlighted as an important component of skill training, as such practices can help therapists tune into and regulate their own in-session reactions and emotions. Several studies have also aimed to address, through training, therapists' anxiety, affect phobia (fear of intense emotional experiences), and the desire to avoid emotionally challenging therapeutic moments. These studies have highlighted the importance of increasing trainees' emotional awareness, helping trainees manage their reactions to client disclosure and emotional expression, and targeting and challenging clinician anxieties and concerns during psychotherapy skill training.

Overall, research suggests that efforts to improve therapist utilization of disclosure elicitation and emotional activation skills must not only provide "how to" training, but also directly address therapists' reservations, fears, and concerns related to disclosure and emotions. This suggests that providing therapists with a training experience that is experiential, includes practice, direct supervision and feedback, and addresses therapists' reservations and anxieties may be an important approach to increase therapist skills in disclosure elicitation and emotional activation. The current study aims to test the effects of an experiential, supervised training approach on therapy trainees' disclosure elicitation and emotional activation skills, and trainees' self-efficacy and affect phobia (fear of emotions), compared to a standard, didactic training approach. It is hypothesized that the experiential training condition will result in greater improvement in performance of the targeted skills and in higher participant ratings of satisfaction with the training compared to the standard training condition. It is also hypothesized that the experiential training condition will result in a greater increase in trainees' self-efficacy and greater decrease in trainees' affect phobia compared to the standard training condition.

ELIGIBILITY:
Inclusion Criteria:

* Graduate students in mental health-related graduate programs (e.g., social work, counseling, and clinical psychology).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Change in targeted therapy skills from baseline to post-training and 1-month follow-up | Immediately Post-Training and 1-month follow-up
  Participant will respond brief pre-recorded videos of actors portraying clients in therapy, and the participant responses will be recorded and coded for skills acquisition using a structured protocol.

SECONDARY OUTCOMES:
Satisfaction with training content and satisfaction with training learning | Immediately Post-Training and 1-month follow-up
  Satisfaction with Training Scale and Satisfaction with Learning Scale (participant ratings of 1 to 6; higher scores indicate higher satisfaction)
Change in self-efficacy from baseline to 1-month follow-up | 1-month follow-up
  Counselor Activity Self-Efficacy Scales; (0 to 9; higher values = higher self-efficacy)
Change in affect phobia from baseline to 1-month follow-up | 1-month follow-up
  Affect Phobia Test; (1 to 5; lower values = higher affect phobia)
Change in anxiety from baseline to 1-month follow-up | 1-month follow-up
  PROMIS Anxiety Scale; (1 to 5; higher values = greater anxiety)
Change in depression from baseline to 1-month follow-up | 1-month follow-up
  PROMIS Depression Scale; (1 to 5; higher values = greater depression)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Lumley, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University Department of Psychology, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yamin JB, Cannoy CN, Gibbins KM, Krohner S, Rapport LJ, Trentacosta CJ, Zeman LL, Lumley MA. Experiential training of mental health graduate students in emotional processing skills: A randomized, controlled trial. Psychotherapy (Chic). 2023 Dec;60(4):512-524. doi: 10.1037/pst0000495. Epub 2023 Jun 29. PMID 37384434